CLINICAL TRIAL: NCT01133782
Title: Clinical Application of PCR-based Diagnosis of Community-onset Viral Respiratory Infections.
Acronym: luftvagsPCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Strama - the Swedish strategic programme against antibiotic resistance. (Unknown); Capio Research Foundation (Other)
Responsible Party: Johan Westin, University of Gothenburg, Dept of Infectious Diseases/Clinical Virology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: luftvagsPCR-01
Record Dates: First submitted 2010-05-28; First posted 2010-05-31 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2006-10

CONDITIONS: Acute Respiratory Tract Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid result (Experimental): Result of diagnostic PCR panel provided the following day
  Interventions: Procedure: Access to diagnostic test
- Delayed result (No Intervention): Result of dagnostic PCR panel provided within 10+/-2 days at follow-up visit.

INTERVENTIONS:
Procedure: Access to diagnostic test — Randomization to receive a result of diagostic procedure the following day.
  Arms: Rapid result

SUMMARY:
Viral respiratory infections are common worldwide. It has been suggested that nucleic acid amplification tests, enabling a rapid etiologic diagnosis, may be useful in reducing antibiotic prescriptions rates. The objective of this study was to evaluate if access to a multiplex real-time PCR method would have an impact on antibiotic prescriptions for acute respiratory tract infections (ARTIs), in primary care. Adult patients with respiratory tract infections will be prospectively included. Nasopharyngeal and throat swabs will be analyzed with a multiplex real-time PCR method, targeting 13 viruses and two bacteria. Samples will be collected during the winter season (October-April). Patients will be open-label randomised to receive a rapid result (the following day) or a delayed result (after 10+/-2 days). The investigators are planning to include approximately 400 patients. Prescription of antibiotics will be measured at initial visit as well as at a follow-up visit 10+/-2 days later. Primary endpoint is antibiotic prescription in the acute phase (initial visit) and secondary endpoint antibiotic treatment (ongoing or initiated) at follow-up visit. The hypohesis is that access to a method with the ability of providing a rapid etiologic diagnosis of respiratory infections will affect the use of antibiotics in outpatient care of adult patients with ARTI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* At least two of the following symptoms: coryza, congestion, sneezing, sore throat, odynophagi, cough, chest pain, shortness of breath or fever for which teh physician found no other explanation.
* Symptom duration of less than 14 days

Exclusion Criteria:

* >14 days of symptoms
* confirmed bacterial infection
* Hospital acquired infection (>3days in hospital)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Antibiotic treatment prescriped at initial visit | Within 2 days of initial visit
  Antibiotic prescriptions are measured as an outcome of the diagnostic procedure tested.

SECONDARY OUTCOMES:
Antibiotic treatment prescribed or reported at follow-up visit | 10+/-2 days
  Antibiotic prescriptions at follow visit are measured as an outcome of the diagnostic procedure tested.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Brittain-Long R, Westin J, Olofsson S, Lindh M, Andersson LM. Access to a polymerase chain reaction assay method targeting 13 respiratory viruses can reduce antibiotics: a randomised, controlled trial. BMC Med. 2011 Apr 26;9:44. doi: 10.1186/1741-7015-9-44. PMID 21521505